CLINICAL TRIAL: NCT05611710
Title: Anakinra for Dengue Patients With Hyperinflammation - a Randomized Double-blind Placebo-controlled Trial
Brief Title: Anakinra in Dengue With Hyperinflammation ( AnaDen )
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 60DX; 223004/Z/21/Z (Other Grant/Funding Number: The Wellcome Trust)
Record Dates: First submitted 2022-10-19; First posted 2022-11-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Dengue; Dengue With Warning Signs; Severe Dengue; Anakinra; Immuno-modulation; Anti-inflammatory Agents; Macrophage Activation Syndrome; Hyperinflammatory Syndrome; Cytokine Storm
Keywords: Dengue; Hyperinflammatory syndrome; Anakinra; Vietnam
MeSH Terms: conditions — Dengue; Severe Dengue; Macrophage Activation Syndrome; Cytokine Release Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blinded, placebo controlled trial of anakinra in patients with dengue with warning signs or severe dengue
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): The control group will be formed of 80 dengue patients with warning signs or severe dengue receiving placebo.
  Interventions: Drug: Placebo
- Anakinra (Experimental): The intervention group will include 80 dengue patients with warning signs or severe dengue receiving anakinra.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Placebo — Drug: Placebo, with visually matched clear syringes
  * Adults (≥16 years) and children (12-16 years, > 50Kg) will receive 2 syringes of placebo via IV route, twice daily for 4 days
  * Children (12-16 years, < 50Kg) will receive no more than 1 syringe of placebo via IV route, twice daily for 4 days
  Arms: Placebo
Drug: Anakinra — Drug: Anakinra
  * Adults (≥16 years) and children (12-16 years, > 50Kg) will receive 200mg of anakinra (2 syringes) via IV route, twice daily for 4 days
  * Children (12-16 years, < 50Kg) will receive 2mg/Kg of anakinra via IV route, twice daily for 4 days (no more than 1 syringe of anakinra, twice daily for 4 days)
  Arms: Anakinra

SUMMARY:
This study aims to evaluate the effect of anakinra in dengue patients with hyperinflammation as compared to placebo

Primary Objective:

To evaluate the efficacy of Anakinra in moderate-severe dengue patients with hyperinflammation.

Secondary Objectives:

* To assess the safety of anakinra therapy in dengue with hyperinflammation
* To assess the effect of anakinra therapy in patients with dengue on physiological, clinical and virological parameters
* To assess the immunomodulation effects of anakinra in dengue
* Immune cell signatures in dengue with and without anakinra
* To assess difference in gene expression between treatment group compared to non-treatment population

DETAILED DESCRIPTION:
This is a randomized double blinded placebo controlled trial investigating the effects of four days of anakinra treatment on dengue patients with hyperinflammatory syndrome. The anakinra/placebo will be given to eligible participants admitted to the Hospital for Tropical Diseases (HTD) in Ho Chi Minh City, Vietnam. 160 dengue patients will be randomly assigned to either anakinra or placebo intervention group to receive treatment for 4 days.

Patients admitted to the HTD with a clinical diagnosis of dengue and at least 1 warning sign(s) or severe dengue to Emergency department / inpatient wards / Intensive Care Units (ICU), will be invited to participate in the trial.

Eligible patients will be invited to participate in the screening phase during which, the collection of clinical information about this acute illness episode as well as some screening tests will be performed, including measurement ferritin, creatinine, pregnancy test (for all females).

- If ferritin level is greater than 2000ng/mL and meet all other inclusion/exclusion criteria, patients will be invited to participate in the randomization phase (second consent), which they will be randomly given either anakinra or placebo intravenous (IV) for four days.

The intervention:

* (i) 200mg bid for four days in adults participants (≥ 16 years) or in children (12-16 years), with weight > 50kg; and
* (ii) 2mg/kg bid for four days in children (12-16 years), with weight < 50Kg.

All patients will be followed up daily at the clinical wards until discharge.

Details of all AEs and SAEs will be recorded on specific forms, together with an assessment as to whether the events are likely to have been related to any treatment received. All SAEs will be reported promptly to the DMC and ECs according to policy. In cases of discontinuation due to AEs, participants will be followed up until the events have resolved or stabilized.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised with a clinical diagnosis of dengue and at least 1 warning sign(s) (see appendix) or severe dengue to Emergency department/inpatient wards/Intensive Care wards (ICU),
* Ferritin levels > 2000ng/mL
* ≥ 12 years of age
* Written informed consent or assent to participate in the study
* Agree to come back for 2 follow up visits around day 30 of illness (maximum 5 weeks) and at 3 months

Exclusion Criteria:

* Pregnancy
* Localizing features suggesting an alternative/additional diagnosis, e.g. pneumonia, sepsis
* Patients taking immunosuppressive drugs or other biologics in last 1 month
* Patients with underlying malignancy or immunosuppression
* Children <12 years
* Have end-stage renal failure (baseline GFR < 30ml/min)
* Being treated for TB
* Taking any drug with significant interaction with anakinra
* The study physician judges that the patient is unlikely to attend follow up visit at around 3-4 weeks after fever onset - e.g. due to long travelling distance from the clinic

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in modified Sequential Organ Failure Assessment score (mSOFA core, modified for limited resource settings and dengue) within 4 days | baseline, up to day 4
  Change in mSOFA score over 4 days after randomization (min score= 0, max score = 24, higher scores mean worse outcomes)

SECONDARY OUTCOMES:
Mortality | Up to day 30
  Number of death up to day 30
Change in modified Sequential Organ Failure Assessment score (mSOFA core, modified for limited resource settings and dengue) at day 7 | baseline, day 7
  Change in mSOFA score at day 7 post randomization (min score= 0, max score = 24, higher scores mean worse outcomes)
Number of days treated in Intensive care unit (ICU) | Up to day 30
  Number of days treated in ICU
Number of days treated in hospital | Up to day 30
  Number of days treated in hospital
Number of participants with Serious Adverse Events (SAEs) | Day 1-5 and Day 6-30
  Number of participants having SAEs within 2 time-periods, 1- 5 days and 6-30 days
Number of Adverse Events (AEs) per participant | Up to day 30
  Number of AEs per individual
Change in Platelets count | Up to day 5, at day 30
  Change in blood levels (Platelets) over 5 days following randomization and at day 30
Change in neutrophils count | Up to day 5, at day 30
  Change in blood levels (neutrophils) over 5 days following randomization and at day 30
Change of ALT levels | Up to day 5, at day 30
  Change in blood levels (ALT) over 5 days following randomization and at day 30
Change of Ferritin levels | Up to day 5, at day 30
  Change in blood levels (Ferritin) over 5 days following randomization and at day 30
Change of CRP levels | Up to day 5, at day 30
  Change in blood levels (CRP) over 5 days following randomization and at day 30
Time to normalization of blood levels | Up to day 30
  Time to normalization of platelets (defined as >150 x109/l) and neutrophils (>2 x109/l)
Platelet nadir | Up to day 30
  Lowest platelet count recorded during admission
Fever clearance time | Up to day 30
  Time to temperature <37.5 for at least 48 hours
Duration of viraemia | Up to day 30
  Number of days from enrollment to the first undetectable viraemia (negative in qPCR and NS1)
Area under the curve (AUC) of the serial viral load measurements during hospital stay | at discharge (assessed up to day 8)
  AUC of viral load measurements during hospital stay will be reported
Patients' quality of life questionnaire score | at discharge (assessed up to day 8) and at day 30
  Patients' quality of life during their hospitalisation will be explored at discharge and day 30 using the EQ-5D questionnaire.

OTHER OUTCOMES:
Change in immune cells | Up to day 90
  Phenotyping CD8/4+T and NK cells will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Yacoub, Principal Investigator — University of Oxford, UK
Locations (1):
- Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data of this study may be requested for publication by journals. Sharing anonymised with future similar/suitable studies will be decided by the sponsor, PIs and the authority agency where the data was collected. No identifiable information will be shared with any other person/organisation than authorized in the study.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Background] Simmons CP, Farrar JJ, Nguyen vV, Wills B. Dengue. N Engl J Med. 2012 Apr 12;366(15):1423-32. doi: 10.1056/NEJMra1110265. No abstract available. PMID 22494122
- [Background] Yacoub S, Wills B. Predicting outcome from dengue. BMC Med. 2014 Sep 4;12:147. doi: 10.1186/s12916-014-0147-9. PMID 25259615
- [Background] Whitehorn J, Yacoub S, Anders KL, Macareo LR, Cassetti MC, Nguyen Van VC, Shi PY, Wills B, Simmons CP. Dengue therapeutics, chemoprophylaxis, and allied tools: state of the art and future directions. PLoS Negl Trop Dis. 2014 Aug 28;8(8):e3025. doi: 10.1371/journal.pntd.0003025. eCollection 2014 Aug. PMID 25166493
- [Background] Tam DT, Ngoc TV, Tien NT, Kieu NT, Thuy TT, Thanh LT, Tam CT, Truong NT, Dung NT, Qui PT, Hien TT, Farrar JJ, Simmons CP, Wolbers M, Wills BA. Effects of short-course oral corticosteroid therapy in early dengue infection in Vietnamese patients: a randomized, placebo-controlled trial. Clin Infect Dis. 2012 Nov;55(9):1216-24. doi: 10.1093/cid/cis655. Epub 2012 Aug 3. PMID 22865871
- [Background] McBride A, Mehta P, Rivino L, Ramanan AV, Yacoub S. Targeting hyperinflammation in infection: can we harness the COVID-19 therapeutics momentum to end the dengue drugs drought? Lancet Microbe. 2021 Jul;2(7):e277-e278. doi: 10.1016/S2666-5247(21)00087-2. Epub 2021 Apr 20. No abstract available. PMID 33899037
- [Background] Dinarello CA. The IL-1 family and inflammatory diseases. Clin Exp Rheumatol. 2002 Sep-Oct;20(5 Suppl 27):S1-13. PMID 14989423
- [Background] van de Weg CA, Huits RM, Pannuti CS, Brouns RM, van den Berg RW, van den Ham HJ, Martina BE, Osterhaus AD, Netea MG, Meijers JC, van Gorp EC, Kallas EG. Hyperferritinaemia in dengue virus infected patients is associated with immune activation and coagulation disturbances. PLoS Negl Trop Dis. 2014 Oct 9;8(10):e3214. doi: 10.1371/journal.pntd.0003214. eCollection 2014 Oct. PMID 25299654
- [Background] Slaats J, Ten Oever J, van de Veerdonk FL, Netea MG. IL-1beta/IL-6/CRP and IL-18/ferritin: Distinct Inflammatory Programs in Infections. PLoS Pathog. 2016 Dec 15;12(12):e1005973. doi: 10.1371/journal.ppat.1005973. eCollection 2016 Dec. PMID 27977798
- [Background] Soundravally R, Agieshkumar B, Daisy M, Sherin J, Cleetus CC. Ferritin levels predict severe dengue. Infection. 2015 Feb;43(1):13-9. doi: 10.1007/s15010-014-0683-4. Epub 2014 Oct 30. PMID 25354733
- [Background] Cavalli G, Larcher A, Tomelleri A, Campochiaro C, Della-Torre E, De Luca G, Farina N, Boffini N, Ruggeri A, Poli A, Scarpellini P, Rovere-Querini P, Tresoldi M, Salonia A, Montorsi F, Landoni G, Castagna A, Ciceri F, Zangrillo A, Dagna L. Interleukin-1 and interleukin-6 inhibition compared with standard management in patients with COVID-19 and hyperinflammation: a cohort study. Lancet Rheumatol. 2021 Apr;3(4):e253-e261. doi: 10.1016/S2665-9913(21)00012-6. Epub 2021 Feb 3. PMID 33655218
- [Background] Kyriakoulis KG, Kollias A, Poulakou G, Kyriakoulis IG, Trontzas IP, Charpidou A, Syrigos K. The Effect of Anakinra in Hospitalized Patients with COVID-19: An Updated Systematic Review and Meta-Analysis. J Clin Med. 2021 Sep 28;10(19):4462. doi: 10.3390/jcm10194462. PMID 34640480
- [Background] Rich C, Eriksson D, Dolfi F, Jablonska K, Dabbous F, Nazir J. Patients diagnosed with COVID-19 and treated with anakinra: a real-world study in the USA. Clin Exp Immunol. 2022 Apr 4;207(2):218-226. doi: 10.1093/cei/uxab024. PMID 35020840
- [Background] European Medicines Agency. Kineret 2022 [updated 22DEC2021. Available from: https://www.ema.europa.eu/en/medicines/human/EPAR/kineret
- [Background] Kanitkar T, Richardson C, Scobie A, Ireson A, Singh A, Jacobs M, et al. Fatal primary dengue-induced haemophagocytis lymphohistiocytosis (HLH) in a returning traveller from India treated with anakinra for the first time. Clinical Infection in Practice. 2020;7-8
- [Background] Gallagher P, Chan KR, Rivino L, Yacoub S. The association of obesity and severe dengue: possible pathophysiological mechanisms. J Infect. 2020 Jul;81(1):10-16. doi: 10.1016/j.jinf.2020.04.039. Epub 2020 May 12. PMID 32413364
- [Background] Azeredo EL, De Oliveira-Pinto LM, Zagne SM, Cerqueira DI, Nogueira RM, Kubelka CF. NK cells, displaying early activation, cytotoxicity and adhesion molecules, are associated with mild dengue disease. Clin Exp Immunol. 2006 Feb;143(2):345-56. doi: 10.1111/j.1365-2249.2006.02996.x. PMID 16412060
- [Background] Jordan MB, Hildeman D, Kappler J, Marrack P. An animal model of hemophagocytic lymphohistiocytosis (HLH): CD8+ T cells and interferon gamma are essential for the disorder. Blood. 2004 Aug 1;104(3):735-43. doi: 10.1182/blood-2003-10-3413. Epub 2004 Apr 6. PMID 15069016
- [Background] Martinez FO, Gordon S. The M1 and M2 paradigm of macrophage activation: time for reassessment. F1000Prime Rep. 2014 Mar 3;6:13. doi: 10.12703/P6-13. eCollection 2014. PMID 24669294
- [Background] Yacoub S, Lam PK, Huynh TT, Nguyen Ho HH, Dong Thi HT, Van NT, Lien LT, Ha QNT, Le DHT, Mongkolspaya J, Culshaw A, Yeo TW, Wertheim H, Simmons C, Screaton G, Wills B. Endothelial Nitric Oxide Pathways in the Pathophysiology of Dengue: A Prospective Observational Study. Clin Infect Dis. 2017 Oct 16;65(9):1453-1461. doi: 10.1093/cid/cix567. PMID 28673038
- [Background] Miao Y, Zhu HY, Qiao C, Xia Y, Kong Y, Zou YX, Miao YQ, Chen X, Cao L, Wu W, Liang JH, Wu JZ, Wang L, Fan L, Xu W, Li JY. Pathogenic Gene Mutations or Variants Identified by Targeted Gene Sequencing in Adults With Hemophagocytic Lymphohistiocytosis. Front Immunol. 2019 Mar 7;10:395. doi: 10.3389/fimmu.2019.00395. eCollection 2019. PMID 30899265
- [Background] Khor CC, Chau TN, Pang J, Davila S, Long HT, Ong RT, Dunstan SJ, Wills B, Farrar J, Van Tram T, Gan TT, Binh NT, Tri le T, Lien le B, Tuan NM, Tham NT, Lanh MN, Nguyet NM, Hieu NT, Van N Vinh Chau N, Thuy TT, Tan DE, Sakuntabhai A, Teo YY, Hibberd ML, Simmons CP. Genome-wide association study identifies susceptibility loci for dengue shock syndrome at MICB and PLCE1. Nat Genet. 2011 Oct 16;43(11):1139-41. doi: 10.1038/ng.960. PMID 22001756
- [Background] Tomashek KM, Wills B, See Lum LC, Thomas L, Durbin A, Leo YS, de Bosch N, Rojas E, Hendrickx K, Erpicum M, Agulto L, Jaenisch T, Tissera H, Suntarattiwong P, Collers BA, Wallace D, Schmidt AC, Precioso A, Narvaez F, Thomas SJ, Edelman R, Siqueira JB, Cassetti MC, Dempsey W, Gubler DJ. Development of standard clinical endpoints for use in dengue interventional trials. PLoS Negl Trop Dis. 2018 Oct 4;12(10):e0006497. doi: 10.1371/journal.pntd.0006497. eCollection 2018 Oct. PMID 30286085
- [Background] Vietnam Ministry of Health. Guidelines for Dengue Diagnosis, Treatment and Prevention. 2019
- [Background] European Medicines Agency. Kineret: EPAR - Product Information 2022 [updated 20JUL2022. Available from: https://www.ema.europa.eu/en/documents/product-information/kineret-epar-product-information_en.pdf
- [Background] CORIMUNO-19 Collaborative group. Effect of anakinra versus usual care in adults in hospital with COVID-19 and mild-to-moderate pneumonia (CORIMUNO-ANA-1): a randomised controlled trial. Lancet Respir Med. 2021 Mar;9(3):295-304. doi: 10.1016/S2213-2600(20)30556-7. Epub 2021 Jan 22. PMID 33493450
- [Background] Cavalli G, De Luca G, Campochiaro C, Della-Torre E, Ripa M, Canetti D, Oltolini C, Castiglioni B, Tassan Din C, Boffini N, Tomelleri A, Farina N, Ruggeri A, Rovere-Querini P, Di Lucca G, Martinenghi S, Scotti R, Tresoldi M, Ciceri F, Landoni G, Zangrillo A, Scarpellini P, Dagna L. Interleukin-1 blockade with high-dose anakinra in patients with COVID-19, acute respiratory distress syndrome, and hyperinflammation: a retrospective cohort study. Lancet Rheumatol. 2020 Jun;2(6):e325-e331. doi: 10.1016/S2665-9913(20)30127-2. Epub 2020 May 7. PMID 32501454
- [Background] Shakoory B, Carcillo JA, Chatham WW, Amdur RL, Zhao H, Dinarello CA, Cron RQ, Opal SM. Interleukin-1 Receptor Blockade Is Associated With Reduced Mortality in Sepsis Patients With Features of Macrophage Activation Syndrome: Reanalysis of a Prior Phase III Trial. Crit Care Med. 2016 Feb;44(2):275-81. doi: 10.1097/CCM.0000000000001402. PMID 26584195
- [Background] Mehta P, Cron RQ, Hartwell J, Manson JJ, Tattersall RS. Silencing the cytokine storm: the use of intravenous anakinra in haemophagocytic lymphohistiocytosis or macrophage activation syndrome. Lancet Rheumatol. 2020 Jun;2(6):e358-e367. doi: 10.1016/S2665-9913(20)30096-5. Epub 2020 May 4. PMID 32373790
- [Background] Manson J, Hartwell J. Anakinra in the treatment of secondary haemophagocytic lymphohistiocytosis 2020. Available from: http://www.leedsformulary.nhs.uk/docs/10.1.3AnakinraUCLHguideline.pdf
- [Background] Halyabar O, Chang MH, Schoettler ML, Schwartz MA, Baris EH, Benson LA, Biggs CM, Gorman M, Lehmann L, Lo MS, Nigrovic PA, Platt CD, Priebe GP, Rowe J, Sundel RP, Surana NK, Weinacht KG, Mann A, Yuen JC, Meleedy-Rey P, Starmer A, Banerjee T, Dedeoglu F, Degar BA, Hazen MM, Henderson LA. Calm in the midst of cytokine storm: a collaborative approach to the diagnosis and treatment of hemophagocytic lymphohistiocytosis and macrophage activation syndrome. Pediatr Rheumatol Online J. 2019 Feb 14;17(1):7. doi: 10.1186/s12969-019-0309-6. PMID 30764840
- [Background] Phadke O, Rouster-Stevens K, Giannopoulos H, Chandrakasan S, Prahalad S. Intravenous administration of anakinra in children with macrophage activation syndrome. Pediatr Rheumatol Online J. 2021 Jun 29;19(1):98. doi: 10.1186/s12969-021-00585-3. PMID 34187503
- [Background] Kharazmi AB, Moradi O, Haghighi M, Kouchek M, Manafi-Rasi A, Raoufi M, Shoaei SD, Hadavand F, Nabavi M, Miri MM, Salarian S, Shojaei S, Khalili S, Sistanizad M, Sadeghi S, Karagah A, Asgari S, Jaffaraghaei M, Araghi S. A randomized controlled clinical trial on efficacy and safety of anakinra in patients with severe COVID-19. Immun Inflamm Dis. 2022 Feb;10(2):201-208. doi: 10.1002/iid3.563. Epub 2021 Nov 11. PMID 34762351
- [Background] Monteagudo LA, Boothby A, Gertner E. Continuous Intravenous Anakinra Infusion to Calm the Cytokine Storm in Macrophage Activation Syndrome. ACR Open Rheumatol. 2020 May;2(5):276-282. doi: 10.1002/acr2.11135. Epub 2020 Apr 21. PMID 32267081
- [Background] Kavirayani A, Charlesworth JEG, Segal S, Kelly D, Wilson S, Qureshi A, Blanco E, Weitz J, O'Shea D, Bailey K. The Lazarus effect of very high-dose intravenous anakinra in severe non-familial CNS-HLH. Lancet Rheumatol. 2020 Dec;2(12):e736-e738. doi: 10.1016/S2665-9913(20)30361-1. Epub 2020 Oct 15. No abstract available. PMID 33083789
- [Background] Yang BB, Frazier J, McCabe D, Young JD. Population pharmacokinetics of anakinra in subjects with rheumatoid arthritis. Annals of Rheumatic Diseases2001. p. A459-60
- [Background] Yang BB, Baughman S, Sullivan JT. Pharmacokinetics of anakinra in subjects with different levels of renal function. Clin Pharmacol Ther. 2003 Jul;74(1):85-94. doi: 10.1016/S0009-9236(03)00094-8. PMID 12844139
- [Background] Fisher CJ Jr, Dhainaut JF, Opal SM, Pribble JP, Balk RA, Slotman GJ, Iberti TJ, Rackow EC, Shapiro MJ, Greenman RL, et al. Recombinant human interleukin 1 receptor antagonist in the treatment of patients with sepsis syndrome. Results from a randomized, double-blind, placebo-controlled trial. Phase III rhIL-1ra Sepsis Syndrome Study Group. JAMA. 1994 Jun 15;271(23):1836-43. PMID 8196140
- [Background] Opal SM, Fisher CJ Jr, Dhainaut JF, Vincent JL, Brase R, Lowry SF, Sadoff JC, Slotman GJ, Levy H, Balk RA, Shelly MP, Pribble JP, LaBrecque JF, Lookabaugh J, Donovan H, Dubin H, Baughman R, Norman J, DeMaria E, Matzel K, Abraham E, Seneff M. Confirmatory interleukin-1 receptor antagonist trial in severe sepsis: a phase III, randomized, double-blind, placebo-controlled, multicenter trial. The Interleukin-1 Receptor Antagonist Sepsis Investigator Group. Crit Care Med. 1997 Jul;25(7):1115-24. doi: 10.1097/00003246-199707000-00010. PMID 9233735
- [Derived] Huyen TB, Trieu HT, Vuong NL, Minh Nguyet N, Tam DTH, McBride A, Linh NTM, Thuan DT, Phong NT, Trung TN, Huong NTC, Vien TTD, Duyen HTL, Hoa VTM, Watson J, Geskus R, Tho PV, Kestelyn E, Qui PT, Yacoub S. Anakinra for dengue patients with hyperinflammation: protocol for a randomized double-blind placebo-controlled trial. Wellcome Open Res. 2024 Nov 22;9:689. doi: 10.12688/wellcomeopenres.21017.1. eCollection 2024. PMID 39931105